CLINICAL TRIAL: NCT01309100
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Contact Lens
Brief Title: Product Feasibility of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 672E
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Lens (Experimental): Bausch & Lomb investigational silicone hydrogel lens.
  Interventions: Device: Investigational Lens
- Acuvue Oasys Lens (Active Comparator): Johnson & Johnson Acuvue Oasys contact lens.
  Interventions: Device: Acuvue Oasys Lens
- Air Optix Aqua Lens (Active Comparator): Ciba Vision Air Optix Aqua contact lens.
  Interventions: Device: Air Optix Aqua Lens

INTERVENTIONS:
Device: Investigational Lens — Bausch & Lomb investigational silicone hydrogel lens on a daily wear basis for 1 week.
  Arms: Investigational Lens
Device: Acuvue Oasys Lens — Johnson & Johnson Acuvue Oasys contact lens on a daily wear basis for 1 week.
  Arms: Acuvue Oasys Lens
Device: Air Optix Aqua Lens — Ciba Vision Air Optix Aqua contact lens on a daily wear basis for 1 week.
  Arms: Air Optix Aqua Lens

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of investigational contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Subjects must be myopic and require lens correction

Exclusion Criteria:

* Subjects with any systemic disease affecting ocular health.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or are using any ocular medication.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Vaz, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, bilateral, three-way crossover, subject-masked study conducted at six sites in the United States. The first participant was enrolled 11/8/2010 and last participant exited on 12/23/2010.
Pre-assignment Details: 144 participants were equally randomized to one of six treatment sequences. 142 participants completed the study.
Groups:
- Overall Study: Participants were equally randomized to one of 6 treatment sequences: RD2117-01, Air Optix Aqua, Acuvue Oasys; RD2117-01, Acuvue Oasys, Air Optix Aqua; Air Optix Aqua, RD2117-01, Acuvue Oasys; Air Optix Aqua, Acuvue Oasys, RD2117-01; Acuvue Oasys, RD2117-01, Air Optix Aqua; Acuvue Oasys, Air Optix Aqua, RD2117-01. All participants wore each of the 3 lenses for one week.
Period: Overall Study
Arm/Group | Overall Study
Started | 144
Completed | 142
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Positive Slit lamp finding | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Arm/Group | Overall Study
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 144

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (Investigational vs Air Optix Aqua Lens)
Description: The mean difference in distance high contrast logMAR visual acuity(VA) between the investigational lens (RD2117-01) and the Air Optix Aqua control lens.
Time Frame: 1 week
Population: All eligible, dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Investigational Lens: Bausch & Lomb investigational silicone hydrogel lens (RD2117-01).
  Investigational Lens: Bausch & Lomb investigational silicone hydrogel lens on a daily wear basis for 1 week.
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 143 | 143
Number analyzed (eyes) | 286 | 286
LogMAR
  Baseline | -0.050 (0.116) | -0.060 (0.116)
  1 Week follow-up | -0.034 (0.111) | -0.039 (0.111)

2. Secondary Outcome: Comfort Throughout the Day (Investigational vs Acuvue Oasys Lens)
Description: The mean differences in comfort between the investigational lens (RD2117-01) and the Acuvue Oasys control lens. Comfort was measured on a scale of 0 to 100, with 100 being the most favorable score.
Time Frame: 1 week
Population: 1-Week Follow-up, All Eligible, Dispensed Eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Investigational Lens: Bausch & Lomb investigational silicone hydrogel lens(RD2117-01).
  Investigational Lens: Bausch & Lomb investigational silicone hydrogel lens on a daily wear basis for 1 week.
Arm/Group | Investigational Lens | Acuvue Oasys Lens
Number analyzed (Participants) | 143 | 143
Number analyzed (eyes) | 286 | 286
units on a scale | 80.9 (21.4) | 86.5 (21.4)

3. Primary Outcome: Visual Acuity (Investigational vs Acuvue Oasys Lens)
Description: The mean difference in distance high contrast logMAR visual acuity(VA) between the investigational lens(RD2117-01) and the Acuvue Oasys control lens.
Time Frame: 1 week
Population: All eligible, dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Acuvue Oasys Lens
Number analyzed (Participants) | 143 | 143
Number analyzed (eyes) | 286 | 286
LogMAR
  Baseline | -0.050 (0.113) | -0.048 (0.113)
  1-week follow-up | -0.034 (0.109) | -0.033 (0.109)

4. Secondary Outcome: Comfort Throughout the Day (Investigational vs Air Optix Aqua Lens)
Description: The mean differences in comfort between the investigational lens(RD2117-01) and the Air Optix Aqua control lens. Comfort was measured on a scale of 0 to 100, with 100 being the most favorable score.
Time Frame: 1 week
Population: All eligible, dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 143 | 142
Number analyzed (eyes) | 286 | 284
units on a scale | 80.9 (21.4) | 82.1 (21.4)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/144
Other Adverse Events (participants affected / at risk) | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other